CLINICAL TRIAL: NCT01852565
Title: An Open-Label, Three Period, Single Sequence Study To Determine The Effect Of Repeat Oral Dosing Of Diltiazem On The Pharmacokinetics Of Repeat Oral Dosing Of Darapladib (SB-480848).
Brief Title: Study to Determine the Effect of Repeated Administration of Diltiazem on the Pharmacokinetics of Darapladib (Sb-480848).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115679
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Atherosclerosis
Keywords: CYP3A4; Lp-PLA2; Atherosclerosis; healthy volunteer; Drug interaction
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Darapladib+Diltizem Arm (Experimental): Each subject will receive darapladib EC tablet 160 mg once daily for 10 days followed by darapladib EC tablet 160 mg once daily + diltiazem 240mg once daily for 14 days and then diltiazem 240mg once daily alone for three days
  Interventions: Drug: Darapladib; Drug: Diltiazem

INTERVENTIONS:
Drug: Darapladib — Enteric coated, free base (micronized) white round tablet, 160mg, Oral/repeat dose/10 days (Treatment Period 1), 14 days (Treatment Period 2)
Drug: Diltiazem — Extended release, Blue capsule imprinted with cardizem CD and 240mg on one end, 240 mg, Oral/repeat dose/17 days

SUMMARY:
Darapladib (SB-480848) is a novel, selective, orally active inhibitor of lipoprotein associated phospholipase A2 (Lp-PLA2) currently under clinical development by GlaxoSmithKline as a potential anti-atherosclerosis agent for reduction of major adverse cardiovascular (CV) events in patient populations with chronic coronary heart disease and after an acute coronary syndrome.

This study will determine the effect of repeated administration of diltiazem on the pharmacokinetics of a repeated administration of darapladib. A drug interaction study with a moderate CYP3A4 inhibitor is warranted to provide guidance to prescribing physicians.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG.
* A subject with an alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase or bilirubin laboratory result outside the reference range may be included only if both the Investigator and the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* BMI within the range 19-37 kilogram per square meter (kg/m2) (inclusive).
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter (MlU/ml) and estradiol < 40 picogram/milliliter [(pg/ml) (<147 pmol/L) is confirmatory].
* A female subject is eligible to participate if she is of Child-bearing potential and is abstinent or agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the final follow-up visit.
* A female subject is eligible to participate if she is of Child-bearing potential and has only same-sex partners, when this is her preferred and usual lifestyle.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Single QT duration corrected for heart rate by Fridericia's formula (QTcF) < 450 Millisecond (msec)

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Criteria Based Upon Medical Histories

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, including diltiazem, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Any contraindications for diltiazem administration.
* Any condition that, in the opinion of the investigator, presents undue risk from the study medications, including diltiazem, or procedures.
* Requiring the use of oral or injectable strong Cytochrome P450 (CYP3) A4 inhibitors or use of other CYP3A4 inhibitor/inducers within 14 days prior to dosing.
* History of anaphylaxis, anaphylactoid (resembling anaphylaxis) reactions
* Clinical criteria for diagnosing anaphylaxis or severe allergic response. Criteria Based Upon Diagnostic Assessments
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Pregnant females as determined by positive human chorionic gonadotropin (hCG) test at screening or prior to dosing.

Other Criteria

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Unwillingness or inability to follow the procedures outlines in the protocol.
* Subject is mentally or legally incapacitated.
* Consumption of grapefruit or grapefruit juice within 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
AUC(0-24h) of darapladib | Up to 32 days. (PK samples will be collected on Days 8, 9, 26 and 27 at predose. Day 10 and Day 28 predose and at 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24, 32, 48, 72, and 96 hours post-dose)
  The area under the concentrations-time curve (AUC0-24) from the time of administration of darapladib up to 24 h after administration.
Cmax of darapladib | Up to 32 days. (PK samples will be collected on Days 8, 9, 26 and 27 at predose. Day 10 and Day 28 predose and at 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24, 32, 48, 72, and 96 hours post-dose)
  The maximum concentration (Cmax) was obtained directly from the measured concentration-time curves.

SECONDARY OUTCOMES:
Number of subjects with adverse event (AE). | Up to 70 days.
  AE's will be collected from the start of study treatment to the last follow up.
12-Lead electrocardiogram (ECG) assessment as a measure of safety and tolerability | Up to 42 days. (Screening Day 32 and Follow up [Day 38 to 42]).
  Single 12-lead ECGs will be obtained after the subject has been in a supine position for at least 10 minutes at each timepoint during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcF intervals.
Vital signs assessment as a measure of safety and tolerability | Up to 42 days (Screening, Day -1, 15, 16, 22, 28, 32 and Follow up [Day 38 to 42]).
  Systolic and diastolic blood pressure and pulse rate measurements will be recorded after the subject has been resting in a semi-supine or supine position for at least 10 minutes.
Safety laboratory tests assessment as a measure of safety and tolerability | Up to 42 days (Screening, Day -1, 15, 32 and Follow up [Day 38 to 42]).
  Hematology, clinical chemistry, urinalysis were assessed.
Tmax and t1/2 of darapladib. | Up to 32 days (PK samples will be collected on Days 8, 9, 26 and 27 at predose. Day 10 and Day 28 predose and at 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24, 32, 48, 72, and 96 hours post-dose.
  Tmax is defined as the time required reaching the maximum concentration of the drug in the plasma after its administration. t1/2 is defined as the time taken to reach half the concentration of the drug after administration.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115679 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115679?search=study&search_terms=115679#rs
- Available data/document: Clinical Study Report: 115679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115679 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register